CLINICAL TRIAL: NCT01288469
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Fixed Dose/Dose Regimen, Multicenter Study Evaluating the Efficacy and Safety of SAR236553 When Co-administered With 80 mg of Atorvastatin Over 8 Weeks in Patients With Primary Hypercholesterolemia and LDL-cholesterol ≥ 100 mg/dL (≥2.59 mmol/L) on Atorvastatin 10 mg
Brief Title: Efficacy and Safety Evaluation of Alirocumab (SAR236553/REGN727) When Co-administered With High Dose of Atorvastatin in Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFI11566; U1111-1117-9994 (Other: UTN)
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-01

CONDITIONS: Hypercholesterolemia
Keywords: 10020603
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo + Atorvastatin 80 mg (Placebo Comparator): Placebo (for alirocumab) subcutaneous (SC) administration every 2 weeks (Q2W) in combination with atorvastatin 80 mg orally once daily for 8 weeks.
  Interventions: Drug: Placebo (for alirocumab); Drug: Atorvastatin
- Alirocumab + Atorvastatin 10 mg (Experimental): Alirocumab 150 mg SC administration Q2W in combination with atorvastatin 10 mg orally once daily for 8 weeks.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin; Drug: Placebo (for atorvastatin)
- Alirocumab + Atorvastatin 80 mg (Experimental): Alirocumab 150 mg SC administration Q2W in combination with atorvastatin 80 mg orally once daily for 8 weeks.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin

INTERVENTIONS:
Drug: Alirocumab — One subcutaneous (SC) injection in the abdomen only.
  Other Names: SAR236553; REGN727
  Arms: Alirocumab + Atorvastatin 10 mg; Alirocumab + Atorvastatin 80 mg
Drug: Placebo (for alirocumab) — One SC injection in the abdomen only.
  Arms: Placebo + Atorvastatin 80 mg
Drug: Atorvastatin — Over-encapsulated tablet orally once daily in the evening with dinner.
Drug: Placebo (for atorvastatin) — One over-encapsulated tablet of placebo for atorvastatin orally once daily in the evening with dinner.
  Arms: Alirocumab + Atorvastatin 10 mg

SUMMARY:
Primary Objective:

To evaluate the effect of alirocumab (SAR236553/REGN727) on low-density lipoprotein cholesterol (LDL-C) levels compared with placebo when co-administered with 80 mg of atorvastatin after 8 weeks of treatment in participants with LDL-C ≥ 100mg/dL (≥ 2.59 mmol/L) on atorvastatin 10 mg.

Secondary Objectives:

* To evaluate the effects of alirocumab on other lipid levels in comparison with placebo, when co-administered with 80 mg of atorvastatin after 8 weeks of treatment.
* To evaluate the efficacy of alirocumab when co-administered with a high dose of atorvastatin (80 mg) versus atorvastatin 10 mg.
* To evaluate the safety and tolerability of alirocumab when co-administered with 2 different doses of atorvastatin.
* To evaluate the development of anti-alirocumab antibodies.
* To evaluate the pharmacokinetics of alirocumab.

DETAILED DESCRIPTION:
The duration of study participation depended on the status of the patient at screening:

* For participants receiving atorvastatin 10 mg at stable dose for at least 6 weeks prior to screening, the study participation was to be approximately 17 weeks including a screening period of 1 week, a double-blind treatment period of 8 weeks and a follow-up period of 8 weeks.
* For participants receiving a lipid lowering treatment other than atorvastatin/ or not at stable dose of atorvastatin 10 mg for at least 6 weeks prior to screening, or drug naive participants, the study participation was to be approximately 23 weeks with a screening period of 1 week, a run-in treatment period with atorvastatin 10 mg of 6 weeks, a double-blind treatment period of 8 weeks and a follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion criteria:

- Participants receiving a lipid-lowering treatment other than atorvastatin/ or not at stable dose of atorvastatin 10 mg for at least 6 weeks prior to screening, or drug naive participants with primary hypercholesterolemia if they are likely to have low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL (≥ 2.59 mmol/L) at the end of the 6-week run-in treatment period on atorvastatin therapy

OR

- Participants with primary hypercholesterolemia treated with stable dose of atorvastatin 10 mg for at least 6 weeks prior to screening and likely to have low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL (≥ 2.59 mmol/L) at the screening visit.

Exclusion criteria:

1. LDL-C < 100 mg/dL (< 2.59 mmol/L) at Week -1 (V1):

   * After the run-in period on atorvastatin 10 mg for participants receiving a lipid lowering treatment other than atorvastatin/ or not at stable dose of atorvastatin 10 mg for at least 6 weeks prior to the screening period, or drug naive participants.

   OR
   * At the first visit for participants who are being treated with atorvastatin 10 mg at stable dose for at least 6 weeks prior to screening visit.
2. Participants not previously instructed on a cholesterol-lowering diet.
3. Participants with type 1 diabetes.
4. Participants with type 2 diabetes treated with insulin.
5. Participants with type 2 diabetes and with an HbA1c ≥ 8.5% at screening visit (considered poorly controlled).
6. Laboratory findings measured before randomization:

   * Triglycerides (TG) > 350 mg/dL (> 3.95 mmol/L) at screening visit.
   * Positive serum or urine pregnancy test in females of childbearing potential.
7. Pregnant or breast-feeding women.
8. Women of childbearing potential with no effective contraceptive method.

The above information is not intended to contain all considerations relevant to a Participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- United States (20):
  - Investigational Site Number 840616, Mesa, Arizona
  - Investigational Site Number 840601, Tucson, Arizona
  - Investigational Site Number 840610, Los Angeles, California
  - Investigational Site Number 840608, Newport Beach, California
  - Investigational Site Number 840603, Doral, Florida
  - Investigational Site Number 840611, Jacksonville, Florida
  - Investigational Site Number 840618, Jupiter, Florida
  - Investigational Site Number 840612, Miami, Florida
  - Investigational Site Number 840614, Miami, Florida
  - Investigational Site Number 840607, St. Petersburg, Florida
  - Investigational Site Number 840605, Chicago, Illinois
  - Investigational Site Number 840619, Chicago, Illinois
  - Investigational Site Number 840604, Edison, New Jersey
  - Investigational Site Number 840606, Rochester, New York
  - Investigational Site Number 840615, Cincinnati, Ohio
  - Investigational Site Number 840617, Cincinnati, Ohio
  - Investigational Site Number 840602, Eugene, Oregon
  - Investigational Site Number 840621, Richmond, Virginia
  - Investigational Site Number 840609, Olympia, Washington
  - Investigational Site Number 840613, Oregon, Wisconsin

REFERENCES:
- [Result] Roth EM, McKenney JM, Hanotin C, Asset G, Stein EA. Atorvastatin with or without an antibody to PCSK9 in primary hypercholesterolemia. N Engl J Med. 2012 Nov 15;367(20):1891-900. doi: 10.1056/NEJMoa1201832. Epub 2012 Oct 31. PMID 23113833
- [Result] Gaudet D, Kereiakes DJ, McKenney JM, Roth EM, Hanotin C, Gipe D, Du Y, Ferrand AC, Ginsberg HN, Stein EA. Effect of alirocumab, a monoclonal proprotein convertase subtilisin/kexin 9 antibody, on lipoprotein(a) concentrations (a pooled analysis of 150 mg every two weeks dosing from phase 2 trials). Am J Cardiol. 2014 Sep 1;114(5):711-5. doi: 10.1016/j.amjcard.2014.05.060. Epub 2014 Jun 18. PMID 25060413
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Toth PP, Hamon SC, Jones SR, Martin SS, Joshi PH, Kulkarni KR, Banerjee P, Hanotin C, Roth EM, McKenney JM. Effect of alirocumab on specific lipoprotein non-high-density lipoprotein cholesterol and subfractions as measured by the vertical auto profile method: analysis of 3 randomized trials versus placebo. Lipids Health Dis. 2016 Feb 13;15:28. doi: 10.1186/s12944-016-0197-4. PMID 26872608

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 20 centers in the United States of America. Overall, 214 participants were screened between January 2011 and April 2011. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:1:1 ratio after confirmation of selection criteria. 92 participants were randomized.
Groups:
- Placebo + Atorvastatin 80 mg: Placebo (for alirocumab) subcutaneous (SC) injection every two weeks (Q2W) in combination with atorvastatin 80 mg orally once daily for 8 weeks.
- Alirocumab + Atorvastatin 10 mg: Alirocumab 150 mg SC injection Q2W in combination with atorvastatin 10 mg orally once daily for 8 weeks.
- Alirocumab + Atorvastatin 80 mg: Alirocumab 150 mg SC injection Q2W in combination with atorvastatin 80 mg orally once daily for 8 weeks.
Period: Overall Study
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Started | 31 (Randomized) | 31 (Randomized) | 30 (Randomized)
Treated | 31 | 31 | 30
Completed | 24 | 28 | 28
Not Completed | 7 | 3 | 2
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Poor compliance to protocol | 0 | 1 | 0
Not completed — Participant Moved | 1 | 0 | 0
Not completed — Consent withdrawn by subject | 1 | 1 | 1
Not completed — Exclusion criteria finally met | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo + Atorvastatin 80 mg: Placebo (for alirocumab) SC injection Q2W in combination with atorvastatin 80 mg orally once daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg | Total
Number analyzed (Participants) | 31 | 31 | 30 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (10.3) | 57.9 (10.0) | 57.6 (9.3) | 56.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 20 | 55
  Male | 13 | 14 | 10 | 37
Low-Density Lipoprotein Cholesterol (LDL-C) in mmol/L [Mean (Standard Deviation); unit: mmol/L] | 3.138 (0.469) | 3.101 (0.402) | 3.288 (0.564) | 3.174 (0.484)
LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] | 121.2 (18.1) | 119.7 (15.5) | 126.9 (21.8) | 122.6 (18.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 8 - On-treatment Analysis
Description: Calculated LDL-C values were obtained using the Friedewald formula. Baseline adjusted least squares (LS) means and standard errors were estimated using an analysis of covariance (ANCOVA) model including available post-baseline data on treatment from first investigational product (IP) injection up to 21 days after last IP injection (on-treatment analysis). Missing Week 8 data were imputed by last observation carried forward [LOCF] method.
Time Frame: From Baseline to Week 8 (LOCF)
Population: Modified Intent-To-Treat (mITT) population: all randomized and treated participants with one baseline and at least one post-baseline calculated LDL-C value on-treatment.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Number analyzed (Participants) | 29 | 29 | 30
percent change | -17.3 (3.5) | -66.2 (3.5) | -73.2 (3.5)
Statistical Analysis 1: Comparison: Placebo + Atorvastatin 80 mg vs Alirocumab + Atorvastatin 80 mg; Throughout the ANCOVA model, the Alirocumab + atorvastatin 80 mg group was compared to the placebo + atorvastatin 80 mg group using appropriate contrast and the 95% confidence interval (CI) of the difference was provided; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤0.05; LS Mean Difference = -55.82, 95% CI 2-sided [-65.62 to -46.03] — Alirocumab vs. placebo

2. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C (mmol/L) at Week 8 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From baseline to Week 8 (LOCF)
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Number analyzed (Participants) | 29 | 29 | 30
mmol/L | -0.56 (0.11) | -2.09 (0.11) | -2.31 (0.11)

3. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C (mg/dL) at Week 8 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From baseline to Week 8 (LOCF)
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Number analyzed (Participants) | 29 | 29 | 30
mg/dL | -21.5 (4.2) | -80.7 (4.2) | -89.3 (4.1)

4. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <100 mg/dL (2.59 mmol/L) and < 70 mg/dL (1.81 mmol/L) at Week 8 - On-treatment Analysis
Time Frame: Week 8 (LOCF)
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Number analyzed (Participants) | 29 | 29 | 30
percentage of participants
  LDL-C < 100 mg/dL (2.59 mmol/L) | 51.7 | 100.0 | 100.0
  LDL-C < 70 mg/dL (1.81 mmol/L) | 17.2 | 96.6 | 90.0

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol, Fasting Triglycerides, Non-high-Density Lipoprotein Cholesterol (Non-HDL-C), Apolipoprotein B (Apo-B) and Lipoprotein(a) at Week 8 - On-treatment Analysis
Description: Since the assumptions of normal distribution and equality of variances were not verified for the lipid parameters, percent changes were expressed as median (interquartile range).
Time Frame: From baseline to Week 8 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post-baseline on treatment value for lipid parameters analyzed. Here, n signifies number of participants analysed for each lipid parameter.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Number analyzed (Participants) | 29 | 29 | 30
percent change
  Total Cholesterol (n=29, 29, 30) | -16.6 [-25.1 to -3.2] | -40.5 [-44.8 to -36.0] | -47.2 [-51.5 to -37.8]
  Fasting Triglycerides (n=29, 29, 30) | -11.9 [-30.4 to 14.3] | -4.0 [-30.5 to 17.4] | -24.7 [-40.3 to -4.4]
  Non-HDL-C (n= 29, 29, 30) | -22.3 [-31.4 to -3.7] | -58.3 [-63.9 to -50.2] | -63.9 [-73.9 to -56.1]
  Apo-B (n = 29, 28, 29) | -12.0 [-23.6 to -3.5] | -54.4 [-60.2 to -48.3] | -58.0 [-67.1 to -46.1]
  Lipoprotein(a) (n= 29, 28, 29) | -2.7 [-19.5 to 16.7] | -34.7 [-50.0 to -24.7] | -31.0 [-50.0 to -15.4]

6. Secondary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) at Week 8 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: From Baseline to Week 8 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post-baseline on treatment HDL-C value.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Number analyzed (Participants) | 29 | 29 | 30
percent change | -3.6 (2.3) | 2.6 (2.3) | 5.8 (2.3)

7. Secondary Outcome: Absolute Change in the Ratio Apolipoprotein B/Apolipoprotein A-1 (ApoB/ApoA-1) From Baseline to Week 8 - On-treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA as for primary endpoint.
Time Frame: From Baseline to Week 8 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post-baseline on treatment value for lipid parameter analyzed
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Placebo + Atorvastatin 80 mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Number analyzed (Participants) | 29 | 28 | 29
ratio | -0.03 [-0.12 to 0.08] | -0.34 [-0.44 to -0.27] | -0.36 [-0.40 to -0.29]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 16) regardless of seriousness or relationship to investigational medicianal product (IMP).
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'treatment emergent period' (the time from the first dose to the last dose of IMP + 70 days). Safety population: participants received at least one dose or partial dose of IMP.
Groups:
- Placebo + Atorvastatin 80mg: Placebo (for alirocumab) SC injection Q2W in combination with atorvastatin 80 mg orally once daily for 8 weeks.
Arm/Group | Placebo + Atorvastatin 80mg | Alirocumab + Atorvastatin 10 mg | Alirocumab + Atorvastatin 80 mg
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 1/30
Other Adverse Events (participants affected / at risk) | 13/31 | 4/31 | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Atorvastatin 80mg (N=31) | Alirocumab + Atorvastatin 10 mg (N=31) | Alirocumab + Atorvastatin 80 mg (N=30)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Atorvastatin 80mg (N=31) | Alirocumab + Atorvastatin 10 mg (N=31) | Alirocumab + Atorvastatin 80 mg (N=30)
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 2 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1
Injection site pruritus (General disorders) | 2 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.